CLINICAL TRIAL: NCT07277244
Title: Low-Intensity Mechanical Ventilation in the Operating Room: a Pilot Study
Acronym: VIOLET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Maximilian S Schaefer, Associate Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P000986
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Robotic Surgery; Post Operative Pulmonary Complications
Keywords: Lung protective ventilation; Electric Impedance Tomography (EIT)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): A guided standard of care protocol will be applied in the control group. This includes a PEEP of 5 cmH₂O, with adjustment by the anesthesia provider if SpO₂ falls below 96% or whenever deemed clinically necessary, a tidal volume of 6-10 mL/kg predicted body weight, and a respiratory rate adjusted to maintain end-tidal CO₂ between 35 and 45 mmHg throughout anesthesia. FiO₂ will be set to 100% during the washout phase at the end of surgery to limit resorption atelectasis.
- Intervention (Experimental): A bundle of protective low-intensity mechanical ventilation strategies will be applied throughout the procedure. All interventions consist of modification of ventilator settings.
  Interventions: Other: Low Intensity Mechanical Ventilation

INTERVENTIONS:
Other: Low Intensity Mechanical Ventilation — A bundle of protective low-intensity mechanical ventilation strategies will be applied throughout the procedure:
  1. Recruitment maneuver
  2. Tidal volume set to 8 ml/kg predicted body weight (PBW) and stepwise adjustment to achieve a driving pressure (Plateau pressure - PEEP) < 13 cmH2O with a minimum tidal volume of 5ml/kg PBW
  3. Respiratory rate adjustment to maintain a target end-tidal carbon dioxide concentration (etCO₂) between 45 and 55 mmHg.
  4. Reassessment and adaptation after Trendelenburg positioning and pneumoperitoneum.
  5. Re-adjustment of Tidal Volume and PEEP ventilator settings to (2.) after exsufflation and return to the supine position. FiO₂ set to 70% during the washout phase of the inhalational anesthetic until extubation.
  Arms: Intervention

SUMMARY:
The aim of the study is to assess whether a bundle of protective low-intensity mechanical ventilation interventions reduces perioperative atelectasis and postoperative pulmonary complications, compared with standard care in a robot-assisted surgical setting. The feasibility of this ventilation bundle will also be assessed.

DETAILED DESCRIPTION:
The investigators hypothesize that protective low-intensity mechanical ventilation during robot-assisted surgery reduces perioperative atelectasis and postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective intra-abdominal or pelvic robot-assisted surgery with a planned duration of at least 2 hours, under general anesthesia with planned extubation at the end of the procedure

Exclusion Criteria:

* Known pregnancy
* Pre-existing intubation or tracheostomy
* Contraindications for esophageal manometry: severe midface trauma or recent nasal surgery, esophageal varices, recent gastric or esophageal surgery
* Contraindications for electrical impedance tomography (EIT): inability to place EIT belt, presence of an active electronic implantable device (e.g., pacemaker, ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
ΔEELV between baseline and after extubation before leaving the operating room. | Perioperative Day 0: From pre-intubation baseline in the operating room (prior to induction of anesthesia) to the first post-extubation EIT assessment (within 10 min after extubation on Day 0).
  Change in end-expiratory lung volume (EELV), measured using electrical impedance tomography between baseline and after extubation before leaving the operating room.

SECONDARY OUTCOMES:
Proportion of patients with postoperative pulmonary complications at day 7 | This secondary outcome will be assessed in the time between day of surgery until 7 days after the day of surgery
  Re-intubation, emergency non-invasive ventilation or pneumonia
Change in right-ventricular systolic function (TAPSE, mm) from pre-intubation baseline to first post-extubation echocardiogram | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, just before extubation
  Right-ventricular systolic function will be assessed by transthoracic echocardiography using tricuspid annular plane systolic excursion (TAPSE, measured in millimeters). TAPSE will be recorded at pre-intubation baseline and at the first postoperative transthoracic echocardiographic examination after extubation. The primary outcome for this measure will be the change in TAPSE (post-extubation minus baseline, mm).
Change in right-ventricular fractional area change (RV-FAC, %) from pre-intubation baseline to first post-extubation echocardiogram | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, just before extubation
  Right-ventricular systolic function will be assessed by transthoracic echocardiography using right-ventricular fractional area change (RV-FAC, expressed as percentage). RV-FAC will be recorded at pre-intubation baseline and at the first postoperative transthoracic echocardiographic examination after extubation. The outcome for this measure will be the change in RV-FAC (post-extubation minus baseline, %).
Change in left ventricular ejection fraction (LVEF, %) from pre-intubation baseline to first post-extubation echocardiogram | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, just before extubation
  Left ventricular systolic function will be assessed by transthoracic echocardiography using left ventricular ejection fraction (LVEF, expressed as percentage). LVEF will be recorded at pre-intubation baseline and at the first postoperative transthoracic echocardiographic examination after extubation. The outcome for this measure will be the change in LVEF (post-extubation minus baseline, %).
Change in estimated pulmonary artery systolic pressure (PASP, mmHg) from pre-intubation baseline to first post-extubation echocardiogram | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, just before extubation
  Pulmonary hemodynamics will be assessed by transthoracic echocardiography using estimated pulmonary artery systolic pressure (PASP, measured in millimeters of mercury). PASP will be recorded at pre-intubation baseline and at the first postoperative transthoracic echocardiographic examination after extubation. The outcome for this measure will be the change in PASP (post-extubation minus baseline, mmHg)
Recruitment rate | Day 0
  Proportion of patients enrolled in the study-defined as those who provided acceptance and signed informed consent-relative to all patients approached.
Intervention deliverability | From intubation to extubation at Day 0
  proportion of patients in the intervention arm in whom the full bundle of protective low-intensity ventilation strategies is delivered as planned across all predefined intraoperative phases.
EELV | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation, after extubation, after PACU admission and 60min after PACU admission
  End-expiratory lung volume measured by Electrical Impedance Tomography in mL
COV | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation, after extubation, after PACU admission and 60min after PACU admission
  Center of ventilation measured by Electrical Impedance Tomography in percentage
RVDI | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation, after extubation, after PACU admission and 60min after PACU admission
  Regional ventilation delay inhomogeneity measured by Electrical Impedance Tomography (unitless)
GI | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation, after extubation, after PACU admission and 60min after PACU admission
  Global inhomogeneity index measured by Electrical Impedance Tomography (unitless)
Dorsal ROI | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation, after extubation, after PACU admission and 60min after PACU admission
  Maximum dorsal ratio of impedance measured by Electrical Impedance Tomography (unitless)
EEPL | Perioperative Day 0: after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation
  End-expiratory transpulmonary pressure, calculated as airway pressure minus esophageal pressure (cmH₂O)
EIPL | Perioperative Day 0: after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation
  End-inspiratory transpulmonary pressure, calculated as airway pressure minus esophageal pressure (cmH₂O)
Relationship between body mass index with optimal PEEP | Intraoperative Day 0: after insufflation of pneumoperitoneum and positioning the patient for surgery
  Correlation between BMI (kg/m²) and the optimal positive end-expiratory pressure (PEEP, cmH₂O) determined after pneumoperitoneum insufflation and patient positioning for surgery.
Relationship of the degree of Trendelenburg inclination with optimal PEEP | Intraoperative Day 0: after insufflation of pneumoperitoneum and positioning the patient for surgery
  Correlation between the degree of Trendelenburg inclination (in degree) and the optimal positive end-expiratory pressure (PEEP, cmH₂O) determined after pneumoperitoneum insufflation and patient positioning for surgery.
Relationship of the pneumoperitoneum (insufflation) with optimal PEEP | Intraoperative Day 0: after insufflation of pneumoperitoneum and positioning the patient for surgery
  Correlation between the pneumoperitoneum (insufflation in cmH2O) and the optimal positive end-expiratory pressure (PEEP, cmH₂O) determined after pneumoperitoneum insufflation and patient positioning for surgery.
Intraoperative oxygenation | Perioperative Day 0: before anesthesia, after intubation, after PEEP/TV/RR titration, after insufflation and positioning, after PEEP/TV/RR reassessment, just before extubation, after extubation
  Intraoperative peripheral pulsed oxygen saturation (SpO2)
Postoperative oxygenation | Postoperative Day 0: after PACU admission and 60min after PACU admission
  Postoperative peripheral pulsed oxygen saturation (SpO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schaefer MS, Treschan TA, Gauch J, Neukirchen M, Kienbaum P. Influence of xenon on pulmonary mechanics and lung aeration in patients with healthy lungs. Br J Anaesth. 2018 Jun;120(6):1394-1400. doi: 10.1016/j.bja.2018.02.064. Epub 2018 Apr 13. PMID 29793604
- [Result] Schaefer MS, Wania V, Bastin B, Schmalz U, Kienbaum P, Beiderlinden M, Treschan TA. Electrical impedance tomography during major open upper abdominal surgery: a pilot-study. BMC Anesthesiol. 2014 Jul 5;14:51. doi: 10.1186/1471-2253-14-51. eCollection 2014. PMID 25018668